CLINICAL TRIAL: NCT02163317
Title: Magnetic Resonance Guided Focal Stereotactic Body Radiation Therapy for Localized Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE11813; NCI-2014-01170 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-06-11; First posted 2014-06-13 (Estimated); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Adenocarcinoma of the Prostate; Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Magnetic Resonance Imaging; Menogaril; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (MRI-guided focal SRS) (Experimental): Patients undergo 3 fractions of MRI-guided focal SRS every other day for 1 week. Patients undergo additional MRI scans between the 2nd and 3rd fractionated treatments, at 6 months following the end of radiation therapy, and at 12 and 24 months.
  Interventions: Radiation: stereotactic radiosurgery; Device: magnetic resonance imaging; Other: quality-of-life assessment; Procedure: Serum Prostate Antigen Test; Procedure: Digital Rectal Exam; Behavioral: Expanded Prostate Cancer Index Composite

INTERVENTIONS:
Radiation: stereotactic radiosurgery — Undergo MRI-guided focal SRS
Device: magnetic resonance imaging — Undergo staging MRI with contrast
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Other: quality-of-life assessment — Quality of life scores will be summarized graphically and repeated measures of variance will be conducted to test for changes in scores over time
  Other Names: quality of life assessment; International Prostate Symptom Score / Sexual Health Inventory for Men (IPSS/SHIM) QoL Scores; Health related quality of life (HRQOL)
Procedure: Serum Prostate Antigen Test — Test of the PSA protein in blood. The test will be run every three months for up to two years during the study.
  Other Names: PSA; PSA response
Procedure: Digital Rectal Exam — Exam of rectal health. Performed every three months for up to two years throughout the study.
  Other Names: DRE
Behavioral: Expanded Prostate Cancer Index Composite — This survey measures a patient's function and bother after prostate cancer treatment. It will be analyzed using ANOVA using data collected every 6 months for up to 2 years of the study.
  Other Names: EPIC

SUMMARY:
This pilot clinical trial studies magnetic resonance (MRI)-guided focal stereotactic radiosurgery (SRS) in treating patients with low- or intermediate-risk localized prostate cancer. Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the correlation of histopathology findings in comparison to regions of the prostate reported to be suspicious for harboring tumor burden on multiparametric MRI report/s.

II. Demonstration of the dosimetric and radiobiological advantages of focal stereotactic body radiation therapy (SBRT) versus whole-gland radiation therapy.

III. Evaluation of clinical outcomes in focal SBRT for localized prostate cancer.

OUTLINE:

Patients undergo 3 fractions of MRI-guided focal SRS every other day for 1 week. Patients undergo additional MRI scans between the 2nd and 3rd fractionated treatments, at 6 months following the end of radiation therapy, and at 12 and 24 months.

After completion of study treatment, patients are followed up every 3 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed diagnosis of adenocarcinoma of the prostate
* Patient must have a history/physical examination with digital rectal examination of the prostate within 90 days prior to screening
* Eastern Cooperative Oncology Group (ECOG) performance status must be level 0 or 1 within 60 days prior to registration
* Patient must have a histological evaluation of the prostate biopsy with assignment of a Gleason score to the biopsy material; Gleason scores ≤ 7(3+4)
* Serum creatinine ≤ 1.5 times upper limit of institutional normal (normal: ≤ 1.17 mL/min/1.73 m^2)
* Clinical stage a ≤ T1-T2a (American Joint Committee on Cancer [AJCC] 7th edition)
* Prostate specific antigen (PSA) ≤ 10 ng/mL within 90 days prior to registration; PSA should not be obtained within 10 days after prostate biopsy
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* Patient willing and able to complete the Expanded Prostate Cancer Index Composite (EPIC) questionnaire (baseline, 6, 12 and 24 months post end of radiation therapy)
* Patients must be able to undergo an MRI with contrast
* Bone scan completed within 90 days

Exclusion Criteria:

* Evidence of distant metastases
* Regional lymph node involvement
* Previous radical surgery (prostatectomy), cryosurgery, or high intensity focused ultrasound (HIFU) for prostate cancer
* Previous pelvic irradiation, prostate brachytherapy, or bilateral orchiectomy
* Previous hormonal therapy, such as luteinizing hormone-releasing hormone (LHRH) agonists (e.g., goserelin, leuprolide) or LHRH antagonists (e.g., degarelix), anti-androgens (e.g., flutamide, bicalutamide), estrogens (e.g., diethylstilbestrol [DES]), or surgical castration (orchiectomy)
* Use of finasteride within 30 days prior to registration; PSA should not be obtained prior to 30 days after stopping finasteride
* Use of dutasteride within 90 days prior to registration; PSA should not be obtained prior to 90 days after stopping dutasteride
* Previous or concurrent cytotoxic chemotherapy for prostate cancer
* Severe, active co-morbidity, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
* Transmural myocardial infarction within the last 6 months
* Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
* Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
* Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however, that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol; (patients on Coumadin or other blood thinning agents are eligible for this study)
* Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease and Control (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; protocol-specific requirements may also exclude immuno-compromised patients
* Patients unable to undergo an MRI with contrast

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Number of patients with change in EPIC bowel domain score that was worse than 5 points | Up to 1 year from start of study
  Number of patients with change in EPIC bowel domain score that was worse than 5 points
  A rate for the worse-than-5 point change in bowel score of up to 35% of patients will be considered acceptable, with a rate ≥55% specified as unacceptable
Number of patients with change in EPIC urinary domain score that was worse than 2 points | Up to 1 year from start of study
  Number of patients with change in EPIC urinary domain score that was worse than 2 points
  A rate for the worse-than-2 point change in urinary score of up to 40% will be considered acceptable, with a rate ≥60% unacceptable

SECONDARY OUTCOMES:
PSA response | Up to 2 years from start of study
  Number of patients with PSA failure. Failure occurs when the PSA is first noted to be 2 ng/mL or more than the patient's nadir value post radiation therapy completion
Number of acute gastrointestinal (GI) grade 3+ acute adverse events, evaluated by the Cancer Therapy Evaluation Program (CTEP) active version of the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) | Up to 30 days after the completion of radiation therapy
  Defined as the first occurrence of worst severity of the adverse event =< 30 days after the completion of radiation therapy. Multivariate analysis will be used, and acute rates of GI toxicity will be reported with dose-volume histogram.
Number of acute genitourinary (GU) grade 3+ acute adverse events, evaluated by the CTEP version of the NCI CTCAE | Up to 2 years from start of study
  Defined as the first occurrence of worst severity of the adverse event =< 30 days after the completion of radiation therapy.
Number of late GI grade 3+ acute adverse events, evaluated by the CTEP version of the NCI CTCAE | Up to 2 years from start of study
  Defined as the first occurrence of worst severity of adverse event > 180 days after radiation therapy completion. Multivariate analysis will be used, and acute rates of GI toxicity will be reported with dose-volume histogram.
Number of late GU grade 3+ acute adverse events, evaluated by the CTEP version of the NCI CTCAE | Up to 2 years from start of study
  Defined as the first occurrence of worst severity of adverse event > 180 days after radiation therapy completion.
Number of patients with Disease-free survival | Up to 2 years from start of study
  Defined as From the date of treatment to the date of documentation of disease progression or until the date of death from any cause. Radiographic efficacy will be summarized by calculating Kaplan-Meier curves. Also, 95% confidence intervals will be reported. Descriptive reports of Response Evaluation Criteria in Solid Tumors (RECIST) (1.1) and volumetric findings will be provided.
Time to local progression | Up to 2 years from start of study
  Radiographic efficacy will be summarized by calculating Kaplan-Meier curves. Descriptive reports of RECIST (1.1) and volumetric findings will be provided. Time will be reported in months.
Time to distant failure | Up to 2 years from start of study
  Radiographic efficacy will be summarized by calculating Kaplan-Meier curves. Descriptive reports of RECIST (1.1) and volumetric findings will be provided. Time will be reported in months.

CONTACTS AND LOCATIONS:
Overall Officials: Elisha Fredman, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Fredman E, Traughber B, Kharouta M, Podder T, Lo S, Ponsky L, MacLennan G, Paspulati R, Ellis B, Machtay M, Ellis R. Focal Prostate Stereotactic Body Radiation Therapy With Correlative Pathological and Radiographic-Based Treatment Planning. Front Oncol. 2021 Sep 15;11:744130. doi: 10.3389/fonc.2021.744130. eCollection 2021. PMID 34604088

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/17/NCT02163317/Prot_SAP_002.pdf
  • Informed Consent Form (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT02163317/ICF_001.pdf